CLINICAL TRIAL: NCT02604446
Title: Depot-opioids for Pre- and Postoperative Pain Relief After Primary Knee Arthroplasty. A Double Blinded Randomized Controlled Study. Tapentadol vs Oxycodone vs Placebo
Brief Title: Depot-opioids for Pre- and Postoperative Pain Relief After Primary Knee Arthroplasty.Tapentadol vs Oxycodone vs Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPO-150; 2015-000295-94 (EudraCT Number)
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Joint Diseases
Keywords: Arthroplasty, Replacement, Knee; Analgesics; Administration and dosage; Knee; Postoperational care; Pain management
MeSH Terms: conditions — Joint Diseases; Agnosia | interventions — Tapentadol; Oxycodone; Glucose

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tapentadol (Experimental): depot Tapentadol in addition to usual pain treatment
  Interventions: Drug: Tapentadol; Drug: usual pain treatment
- Oxycodone (Active Comparator): depot Oxycodone in addition to usual pain treatment
  Interventions: Drug: Oxycodone; Drug: usual pain treatment
- Placebo (Placebo Comparator): depot glucose placebo in addition to usual pain treatment.
  Interventions: Drug: Placebo; Drug: usual pain treatment

INTERVENTIONS:
Drug: Tapentadol
  Other Names: Palexia Depot
  Arms: Tapentadol
Drug: Oxycodone
  Other Names: Oxycontin
  Arms: Oxycodone
Drug: Placebo
  Other Names: Glucose
  Arms: Placebo
Drug: usual pain treatment — premedication of Dexamethasone, Paracetamol, Vimovo; postoperative Paracetamol and Vimovo

SUMMARY:
This study will provide knowledge about the use of long-acting opioids for pain relief after primary knee arthroplasty. The investigators will compare depot tapentadol, depot oxycodone and placebo for effect on pain relief and side effects. The three study groups reflect the three different postoperative pain regimens that have been used the last years at St. Olavs Hospital, so investigators know that no patient will receive an inadequate pain treatment. The purpose of the study is to find which of the three treatments that gives the best pain relief with the least amount of side effects. The results will be of use for postoperative pain treatment for knee arthroplasty, but also for other types of major surgery. Similar studies that are not sponsored by pharmaceutical industry have not been published yet.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for knee arthroplasty at St. Olavs University Hospital
* consent in participation in the study

Exclusion Criteria:

* Contraindications for any of the study drugs
* Lactose intolerance
* Known hypersensitivity against any of the additives
* Chronic Obstructive Pulmonary Disease (COPD) grade 3 or 4
* Paralytic ileus
* Known alcohol or medical addiction/abuse
* History of asthma, urticaria or allergic reaction caused by acetyl salicylic acid or other NSAIDs
* Peptic ulcer
* Hemophilia
* Gastrointestinal bleeding
* Cerebrovascular bleeding
* Inflammatory bowel disease (ulcerous colitis, Crohn disease)
* Concomitant use of the following drugs: ACE-inhibitors, AT2-blockers, SSRI, Anti-psychotic drugs, MAO-inhibitors, Atazanavir and Nelfinavir (medicine used for HIV-infection)
* Known kidney failure (creatinin level above reference value)
* Known heart failure (NYHA III-IV)
* Pregnancy
* Women in fertile age with risk of pregnancy
* Nursing women
* operated under general anesthesia without use of spinal anesthesia
* using opioids on a regular basis except users of codeine or tramadol, or known former abuse of opioids
* Cognitive failure or other factors which make follow up impossible (for example language difficulties)
* No cell phone or internet connection at home (making follow up difficult)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-09; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) based on daily numeric rating score (NRS) scale 1-10 for pain by mobilization the first 8 postoperative days | 8 days
  NRS-scores

SECONDARY OUTCOMES:
Pain at rest in the previous 24 hours | 8 days
  NRS-scores 1-10 scale
worst pain in the previous 24 hours | 8 days
  NRS-scores 1-10 scale
quality of sleep in the previous night | 8 days
  NRS-scores 1-10 scale
nausea in the previous 24 hours | 8 days
  NRS-scores 1-10 scale
obstipation in the previous 24 hours | 8 days
  NRS-scores 1-10 scale
dizziness in the previous 24 hours | 8 days
  NRS-scores 1-10 scale
sedation in the previous 24 hours | 8 days
  NRS-scores 1-10 scale
headache | 8 days in the previous 24 hours
  NRS-scores 1-10 scale

CONTACTS AND LOCATIONS:
Overall Officials: Petter Aadahl, md phd, Study Director — St. Olavs Hospital
Locations (1):
- Anestesiavdelingen, St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Rian T, Skogvoll E, Hofstad J, Hovik L, Winther SB, Husby VS, Klaksvik J, Egeberg T, Sand K, Klepstad P, Wik TS. Tapentadol vs oxycodone for postoperative pain treatment the first 7 days after total knee arthroplasty: a randomized clinical trial. Pain. 2021 Feb 1;162(2):396-404. doi: 10.1097/j.pain.0000000000002026. PMID 32773594
- [Derived] Rian T, Sand K, Skogvoll E, Klepstad P, Wik TS. A Web-Based Communication Tool for Postoperative Follow-up and Pain Assessment at Home After Primary Knee Arthroplasty: Feasibility and Usability Study. JMIR Form Res. 2022 Apr 28;6(4):e34543. doi: 10.2196/34543. PMID 35482392